CLINICAL TRIAL: NCT06934031
Title: A Comparative Study of Interpretation Performance of ChatGPT, Google Translate, and UD Talk in Chinese and Japanese Medical Consultation Scenarios: Contexts of Cardiopulmonary Disease Consultation
Brief Title: Interpretation Performance in Chinese and Japanese Medical Consultation Scenarios
Status: Completed | Type: Observational
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Assistant Professor, Fu Jen Catholic University
Other Study IDs: FJUH113419
Record Dates: First submitted 2025-03-31; First posted 2025-04-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Outpatients; Cardiology; Pulmonology
Keywords: Language barriers; medical communication; medical interpretation; cardiopulmonary disease; translation software
MeSH Terms: conditions — Pulmonary Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: translation software — ChatGPT, Google Translate, and UD talk

SUMMARY:
This study aims to compare the translation and interpretation performance of ChatGPT, Google Translate(GT),and UD Talk in cardiopulmonary consultations and analyze their effectiveness in addressing language barriers.The investigators hypothesize that ChatGPT and UD Talk will outperform GT in terms of accuracy and error rates.

DETAILED DESCRIPTION:
Background： Language barriers in healthcare have a significant impact on patient safety, health outcomes, and the quality of healthcare services. With the increase in global migration, more patients are facing language challenges in foreign healthcare systems. Literature shows that providing professional interpretation services significantly improves patient satisfaction and communication quality. However, due to the high usage of ad-hoc interpreters and the shortage of professional interpreters, clinical communication quality has declined.

Study Design： This is a one-year, single-center, prospective observational study. Methods： The study will be conducted in the cardiology and pulmonology outpatient clinics at Fu Jen University Hospital. A total of 20 cardiopulmonary disease patients will be enrolled, withtheir consultation sessions recorded and transcribed into Chinese. The study will compare the three tools' performance in terms of semantic accuracy, error types, and severity, and analyze their feasibility in clinical practice. Further analysis will involve satisfaction surveys from both professional interpreters and non-native speakers living in Taiwan. The translation results will be evaluated for accuracy and error rates by 8 professional medical interpreters, with a satisfaction survey completed by a total of 14 non-experts. The evaluation tool will be based on the assessment rubrics from the National Accreditation Authority for Translators and Interpreters.

Effect： It is expected that ChatGPT and UD Talk will show better translation accuracy and interpretation quality compared to GT. UD Talk is anticipated to perform better than the other two tools in real-time interpretation. The study results will provide valuable insights for future medical interpretation training and clinical applications.

ELIGIBILITY:
First part

Inclusion Criteria:

* Age over 18 years
* Patients visiting the Cardiology or Pulmonology Department at Fu Jen Catholic University Hospital from December 2024 to November 2025

Exclusion Criteria:

* Patients unable to communicate effectively as assessed by the physician
* Refusal to participate in the study

Second part

Inclusion Criteria:

* Age over 18 years
* Completed the Japanese-Chinese medical interpretation training course and has at least two years of clinical experience

Exclusion Criteria:

* Refusal to participate in the study

Third part

Inclusion Criteria:

* Age over 18 years
* Non-native Chinese-speaking Japanese residents who have lived in Taiwan for at least two years

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First part
  * Patients visiting the Cardiology or Pulmonology Department
  Second part
  * Has completed Japanese-Chinese medical interpretation training and has clinical experience
  Third part
  * Non-native Chinese-speaking Japanese residents
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Translation Assessment Scale Score | 4 months
  6-point Likert scale, with 5 representing the highest score and 0 representing the lowest.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No